CLINICAL TRIAL: NCT03419286
Title: Retrospective Study of Cases of Small Cell Lung Cancer (SCLC) That Appeared During Treatment of Another Lung Carcinoma With or Without Oncogenic Activation (TransCPC)
Brief Title: Transformation Into Small Cell Lung Cancer : a Mode of Resistance to Treatment
Acronym: TransCPC
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC16.053
Record Dates: First submitted 2018-01-18; First posted 2018-02-01 (Actual); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- EGFR MUTATED: patient with lung cancer with EGFR mutation before transformation into small cell lung cancer
- EGFR NON MUTATED: patient with lung cancer without driver oncogenic before transformation into small cell lung cancer

SUMMARY:
The discovery of oncogenic mutations and the use of targeted therapies have transformed the management of certain tumors. Thus 12 to 15% of bronchial adenocarcinomas (AD) carry mutations of EGFR and receive from the first line inhibitors of this kinase (ITK). Despite spectacular results, relapse and resistance are quasi-general phenomena. In most known cases, EGFR-TKI resistance mechanisms involve secondary mutations of EGFR or the activation of alternative oncogenic pathways. However, in 5 to 15% of patients, resistance is manifested by the emergence of a small cell carcinoma (CPC), a cancer of neuroendocrine origin very different from AD by its cellular, molecular and epidemiological characteristics. This phenotypic transformation is an almost unique phenomenon in oncology and its molecular bases are not understood. To study this phenomenon, a Franco-Italian network was established that documented and collected cases of this rare tumor. This series is the subject of detailed anatomopathological, clinical and therapeutic documentation. This project aims to investigate the exome of one or more matched lesion regions to evaluate the evolutionary processes leading from the initial AD to the relapsing CPC. These results will guide future research on predictive markers of relapse and their targeted treatment.

DETAILED DESCRIPTION:
An international multicentric retrospective collection of cases was performed between 2005 and 2017. A global e-mailing to a network of thoracic oncology centers in France and Italy called for the selection of retrospective cases. Consecutive non small cell lung cancer (NSCLC) patients with stage III or IV EGFR NSCLC with or without initial EGFR mutation with a secondary transformation to small cell lung cancer (SCLC) in participating centers in France and Italy were included. Patients with a previous history of SCLC or neuroendocrine tumor of the lung were excluded as well as patients with combined Small cell/ Non-small cell lung cancer on the initial pathology sample.

Study ethics approval was obtained on December 8th of 2015 (CECIC Rhône-Alpes-Auvergne, Clermont-Ferrand, IRB 5891). Anonymized data were collected at each center then centrally analyzed at the Albert Bonniot Institute, Inserm U 823, Grenoble Alpes University, in Grenoble, France.

The primary objective of this study was to analyze survival data after transformation to SCLC. The secondary objectives were to define: the epidemiological characteristics at the time of diagnosis of NSCLC, the histomolecular characteristics at the time of diagnosis of NSCLC and at the time of diagnosis of SCLC; the clinical characteristics at the time of diagnosis of NSCLC and SCLC and the treatment characteristics before and after transformation from NSCLC to SCLC.

All identified cases will be analyzed. This concerns about sixty two patients because the transformation into small cell lung cancer is a rare mechanism of resistance, it is for this reason that all the cases will be included in order to obtain the most exhaustive data possible.

Continuous variables were described as median (25%-75% interquartile range [IQR]) and categorical variables as number (%). Associations between categorical variables were compared using the chi-2 test or Fisher's exact test and those between continuous variables using the Wilcoxon test. Patients were followed until November of 2017. Overall survival (OS) is the time from the initial diagnosis of lung cancer to death and survival after SCLC transformation is from the rebiopsy to death. Kaplan-Meier plots of survival curves were compared between groups using the log-rank test. All tests were two-sided, and P values <0.05 were considered statistically significant. All statistical analyses were performed using SAS 9.3 (SAS Institute, Cary, NC, USA).

ELIGIBILITY:
Inclusion Criteria:

* Patient with no history of small cell cancer or Neuroendocrine cancer
* Patients with non-small cell lung cancer at baseline, stage IIIB or IV
* Transformation during treatment of non small cell lung cancer, in small cell cancer proven by biopsy

Exclusion Criteria:

* History of small cell cancer or Neuroendocrine cancer
* Absence of histological evidence of the transformation into small cell lung cancer after treatment of non small cell lung cancer
* Patients with non-small cell lung cancer at initial biopsy, stage I, II, IIIA

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All cases diagnosed between 2005 to 2017 in France and in Italy who respond at the eligibility criteria were included. they are patients with non small cell lung cancer with or without EGFR mutation at the initial diagnosis transformed into small cell lung cancer during treatment of non small cell lung cancer
Sampling Method: Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
survival time after transformation to small cell lung cancer (SCLC) | 2005 to 2017
  months of survival after transformation into small cell lung cancer

SECONDARY OUTCOMES:
time from initial diagnosis of non small cell lung cancer (NSCLC) to small cell lung cancer transformation | 2005 to 2017
  median of months between initial diagnosis of non small cell lung cancer and small cell lung cancer transformation
histology type at the time of diagnosis of NSCLC and at the time of diagnosis of small cell lung cancer (SCLC) | 2005 to 2017
  histology on biopsy at the initial diagnosis and at transformation according with OMS classification
type of specific treatments administered before and after transformation from non small cell lung cancer into small cell lung cancer | 2005 to 2017
  The type of treatment administered before and after SCLC transformation. percentage of patients in each type of specific treatment used
sexe of patients | 2005 to 2017
  sexe female or male in percentage of patients
stage of NSCLC at initial diagnosis | 2005 to 2017
  percentage of patients with stage III and with IV of NSCLC
smocking status at diagnosis initial of non small cell lung cancer | 2005 to 2017
  percentage of patients in never, former or active smokers
type of mutations at the diagnostic initial NSCLC and at transformation | 2005 to 2017
  the mutation on initial biopsy and on biopsy at transformation in SCLC in percentage of patients
treatment lines before transformation into small cell lung cancer (SCLC) | 2005 to 2017
  Median number of lines of treatment for the NSCLC before transformation into SCLC
response rates to first line treatment after transformation into small cell lung cancer | 2005 to 2017
  response rate in percentage of patients after transformation into SCLC according with the RECIST criteria
lines of treatment after transformation into SCLC | 2005 to 2017
  median number of lines of treatment after transformation into SCLC
age of patients | 2005 to 2017
  the median in years at the he diagnosis initial of non small cell lung cancer

CONTACTS AND LOCATIONS:
Overall Officials: Denis Moro-Sibilot, MD-PHD, Principal Investigator — University Hospital, Grenoble

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sequist LV, Waltman BA, Dias-Santagata D, Digumarthy S, Turke AB, Fidias P, Bergethon K, Shaw AT, Gettinger S, Cosper AK, Akhavanfard S, Heist RS, Temel J, Christensen JG, Wain JC, Lynch TJ, Vernovsky K, Mark EJ, Lanuti M, Iafrate AJ, Mino-Kenudson M, Engelman JA. Genotypic and histological evolution of lung cancers acquiring resistance to EGFR inhibitors. Sci Transl Med. 2011 Mar 23;3(75):75ra26. doi: 10.1126/scitranslmed.3002003. PMID 21430269
- [Background] Yu HA, Arcila ME, Rekhtman N, Sima CS, Zakowski MF, Pao W, Kris MG, Miller VA, Ladanyi M, Riely GJ. Analysis of tumor specimens at the time of acquired resistance to EGFR-TKI therapy in 155 patients with EGFR-mutant lung cancers. Clin Cancer Res. 2013 Apr 15;19(8):2240-7. doi: 10.1158/1078-0432.CCR-12-2246. Epub 2013 Mar 7. PMID 23470965
- [Background] Niederst MJ, Sequist LV, Poirier JT, Mermel CH, Lockerman EL, Garcia AR, Katayama R, Costa C, Ross KN, Moran T, Howe E, Fulton LE, Mulvey HE, Bernardo LA, Mohamoud F, Miyoshi N, VanderLaan PA, Costa DB, Janne PA, Borger DR, Ramaswamy S, Shioda T, Iafrate AJ, Getz G, Rudin CM, Mino-Kenudson M, Engelman JA. RB loss in resistant EGFR mutant lung adenocarcinomas that transform to small-cell lung cancer. Nat Commun. 2015 Mar 11;6:6377. doi: 10.1038/ncomms7377. PMID 25758528
- [Background] Oser MG, Niederst MJ, Sequist LV, Engelman JA. Transformation from non-small-cell lung cancer to small-cell lung cancer: molecular drivers and cells of origin. Lancet Oncol. 2015 Apr;16(4):e165-72. doi: 10.1016/S1470-2045(14)71180-5. PMID 25846096
- [Background] Crystal AS, Shaw AT, Sequist LV, Friboulet L, Niederst MJ, Lockerman EL, Frias RL, Gainor JF, Amzallag A, Greninger P, Lee D, Kalsy A, Gomez-Caraballo M, Elamine L, Howe E, Hur W, Lifshits E, Robinson HE, Katayama R, Faber AC, Awad MM, Ramaswamy S, Mino-Kenudson M, Iafrate AJ, Benes CH, Engelman JA. Patient-derived models of acquired resistance can identify effective drug combinations for cancer. Science. 2014 Dec 19;346(6216):1480-6. doi: 10.1126/science.1254721. Epub 2014 Nov 13. PMID 25394791
- [Background] Ross JS, Wang K, Elkadi OR, Tarasen A, Foulke L, Sheehan CE, Otto GA, Palmer G, Yelensky R, Lipson D, Chmielecki J, Ali SM, Elvin J, Morosini D, Miller VA, Stephens PJ. Next-generation sequencing reveals frequent consistent genomic alterations in small cell undifferentiated lung cancer. J Clin Pathol. 2014 Sep;67(9):772-6. doi: 10.1136/jclinpath-2014-202447. PMID 24978188
- [Background] Suda K, Murakami I, Sakai K, Mizuuchi H, Shimizu S, Sato K, Tomizawa K, Tomida S, Yatabe Y, Nishio K, Mitsudomi T. Small cell lung cancer transformation and T790M mutation: complimentary roles in acquired resistance to kinase inhibitors in lung cancer. Sci Rep. 2015 Sep 24;5:14447. doi: 10.1038/srep14447. PMID 26400668
- [Background] Du L, Schageman JJ, Irnov, Girard L, Hammond SM, Minna JD, Gazdar AF, Pertsemlidis A. MicroRNA expression distinguishes SCLC from NSCLC lung tumor cells and suggests a possible pathological relationship between SCLCs and NSCLCs. J Exp Clin Cancer Res. 2010 Jun 17;29(1):75. doi: 10.1186/1756-9966-29-75. PMID 20624269
- [Background] Shoemaker AR, Mitten MJ, Adickes J, Ackler S, Refici M, Ferguson D, Oleksijew A, O'Connor JM, Wang B, Frost DJ, Bauch J, Marsh K, Tahir SK, Yang X, Tse C, Fesik SW, Rosenberg SH, Elmore SW. Activity of the Bcl-2 family inhibitor ABT-263 in a panel of small cell lung cancer xenograft models. Clin Cancer Res. 2008 Jun 1;14(11):3268-77. doi: 10.1158/1078-0432.CCR-07-4622. PMID 18519752
- [Background] Lee JK, Lee J, Kim S, Kim S, Youk J, Park S, An Y, Keam B, Kim DW, Heo DS, Kim YT, Kim JS, Kim SH, Lee JS, Lee SH, Park K, Ku JL, Jeon YK, Chung DH, Park PJ, Kim J, Kim TM, Ju YS. Clonal History and Genetic Predictors of Transformation Into Small-Cell Carcinomas From Lung Adenocarcinomas. J Clin Oncol. 2017 Sep 10;35(26):3065-3074. doi: 10.1200/JCO.2016.71.9096. Epub 2017 May 12. PMID 28498782